CLINICAL TRIAL: NCT04082923
Title: Does Meal Texture Have Different Impact on Glucose Metabolism and Intestinal Hormone Response After Gastric Bypass and Sleeve Gastrectomy Operated Patients?
Brief Title: Effect of Meal Texture on Glucose-metabolism and Gut Hormone Response After Bariatric Surgery
Acronym: Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Nora Elisabeth Hedbäck, MD, principal inverstigator, Hvidovre University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H-19027100
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Glucose Metabolism Disorders; Obesity; Sleeve Gastrectomy; Gastric Bypass; Gut Hormones
MeSH Terms: conditions — Glucose Metabolism Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gastric bypass operated patients (Other): Two test days in a randomized, patient-blinded, cross-over design
  Interventions: Other: Liquid meal; Other: Solid meal
- Gastric sleeve operated patients (Other): Two test days in a randomized, patient-blinded, cross-over design
  Interventions: Other: Liquid meal; Other: Solid meal
- Control arm (Other): Two test days in a randomized, patient-blinded, cross-over design
  Interventions: Other: Liquid meal; Other: Solid meal

INTERVENTIONS:
Other: Liquid meal — Four-hour liquid mixed meal test
Other: Solid meal — Four-hour solid mixed meal test

SUMMARY:
The investigators want to evaluate the difference in glucose metabolism and intestinal hormonal response after a liquid meal versus a solid meal in patients after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* RYGB or SG operation > 12 months prior to inclusion
* Weight stable (± 3 kg during the last month)
* HbA1c < 48 mmol/mol before surgery, and no history of diabetes
* HbA1c < 48 mmol/mol and fasting plasma glucose < 6.1 mmol/l at inclusion

Exclusion Criteria:

* Thyrotoxicosis or inadequately treated hypothyreosis
* Hemoglobin < 6.5 mmol/l at inclusion
* Pregnancy or breast feeding
* Medication affecting the planned examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
GLP-1 response | 240 minutes
  GLP-1 response after a liquid meal test compared to a solid meal test

SECONDARY OUTCOMES:
Difference in gut hormone response after bariatric surgery | 240 minutes

CONTACTS AND LOCATIONS:
Overall Officials: NOra Hedbäck, MD, Principal Investigator — Department of Endocrinology Hvidovre Hospital Denmark
Locations (1):
- Department of Endocrinology, Hvidovre University Hospital, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Hedback N, Hindso M, Bojsen-Moller KN, Linddal AK, Jorgensen NB, Dirksen C, Moller A, Kristiansen VB, Hartmann B, Holst JJ, Svane MS, Madsbad S. Effect of Meal Texture on Postprandial Glucose Excursions and Gut Hormones After Roux-en-Y Gastric Bypass and Sleeve Gastrectomy. Front Nutr. 2022 Apr 29;9:889710. doi: 10.3389/fnut.2022.889710. eCollection 2022. PMID 35571890